CLINICAL TRIAL: NCT07119151
Title: Multicentric Prospective Observational Study of Neodent Implantable Devices of Helix Short System
Status: Not yet recruiting | Type: Observational
Sponsor: Neodent (Industry)
Collaborators: Federal University of Uberlandia (Other); UNESP, Câmpus de Araraquara (Other); Faculdade ILAPEO (Unknown)
Responsible Party: Sponsor
Other Study IDs: CS.O.014
Record Dates: First submitted 2025-07-29; First posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Edentulism; Dental Implant; Atrophy of Edentulous Alveolar Ridge; Atrophy of Edentulous Mandibular Alveolar Ridge; Atrophy of Edentulous Maxillary Alveolar Ridge
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Treatment: Patients with maxillary and mandible atrophy in need of one or more dental implants and who were evaluated as suitable for the installation of Helix Short implants.
  Interventions: Device: Dental Implant

INTERVENTIONS:
Device: Dental Implant — Dental Implant placement and loading.

SUMMARY:
This is a post-market prospective observational study to prospectively collect clinical data to confirm the long-term safety and clinical performance of implants and abutments Helix Short in a daily dental practice setting, by means of success and survival rates of these devices. Additionally, from the collected data, the study aims to identify previously unknown side-effects and monitor the known side-effects and contraindications stated on the IFU, identify and analyze emerging risks on the basis of factual evidence, and ensure the continued acceptability of the benefit-risk ratio with the intent to verify that the intended purpose is correct for all JJGC products involved in the procedure that get in contact with the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with atrophic maxilla and mandible, who need of one or more dental implants with opposing dentition (natural teeth or teeth/implant-supported fixed restorations) and who qualify for placement of Helix Short implants.
* Collaborative patient.
* Patient with opposing dentition (natural teeth or fixed and/or removable restorations)

Exclusion Criteria:

* Contraindication according to the IFU: This product is contraindicated for patients who show signs of allergy or hypersensitivity to the chemical components of titanium. Implants with a length of 4 mm are contraindicated for single and overdenture rehabilitations, and they are contraindicated for total and multiple restorations when not associated with implants with lengths greater than or equal to 5.5 mm.
* Patients with periodontal disease, severe alcohol/tobacco consumption, bruxism, high use of bisphosphonates or proton pump inhibitors (PPI), radiotherapy to the neck and head in the last 3 years, uncontrolled systemic diseases.
* Pregnant patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with atrophic maxilla and mandible, who need of one or more dental implants with opposing dentition (natural teeth or teeth/implant-supported fixed restorations) and who qualify for placement of Helix Short implants.
Sampling Method: Non-Probability Sample
Enrollment: 94 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Implant success rate | From the implant loading to the 36-months of follow-up
  Implant success rate (including survival as one of the criteria for success) of implants at 3 years after implant loading.

SECONDARY OUTCOMES:
Implant survival rate | From the implant loading to the 36-months of follow-up
  Implant survival rate
Prosthetic survival and success rates | From the implant loading to 36-months of follow-up
  Prosthetic results
Change in peri-implant bone level | From the implant loading to 36-months of follow-up
  Evaluating bone loss
Soft tissue assessment - Visible Plaque | From the implant loading to 36-months of follow-up
  Visible plaque index will be calculated for each implant site as the percentages of surfaces (mesial, buccal, distal, lingual) presenting visible plaque.
Evaluation of the crown/implant ratio | From the implant loading to 36-months of follow-up
  Evaluation of the crown/implant ratio
Risk factors for Implant Loss | From the enrollment to 36-months of follow-up
  Risk factors for implant loss will be assessed performing statistical analysis between implants losses and characteristics of these losses (implant and procedures' characteristics).
Type of load and time for final prosthesis | From the implant placement to 36-months of follow-up
  If immediate or late loading.
Patient satisfaction | From the enrollment to 36-months of follow-up.
  Patient satisfaction assessment through (Oral Health Impact Profile-14) questionnaire. It is made of 14 questions to be answered through a set of Likert scale. The final score is calculated based on the answers for each question, and it is ranged from 0 to 56. The highest score indicates a greater negative impact of oral health on a person's well-being. The questions include seven dimensions: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and social disadvantage. The questionnaire will be applied in different times of follow-up during the study.
Clinician satisfaction with all devices used and procedures | From the implant placement to 36-months of follow-up.
  Clinician satisfaction assessment through a questionnaire about implant placement and rehabilitation outcomes, and the answers through a visual analogue scale (VAS) from 1 to 10. The highest scores means better outcome.
Adverse events and residual risks related to the implant, prosthetic component, and prosthesis. | From the enrollment to 36-months of follow-up.
  Monitoring of adverse events, including implant and prothesis loss to evaluate their association with implant's and patient's charactheristics.
Soft tissue assessment - Marginal Bleeding Indexes | From the implant loading to 36-months of follow-up
  Marginal bleeding index will be calculated for each implant site as the percentages of surfaces (mesial, buccal, distal, lingual) presenting marginal bleeding.
Soft tissue assessment - Bleeding on probing | From the implant loading to 36-months of follow-up
  Bleeding on probing will be assessed as present or absent, using a periodontal probe to the bottom of the clinical sulcus, in the buccal surface of each implant site. Bleeding will be considered positive if it occurs within 10 to 15 seconds after probing.
Soft tissue assessment - Keratinized gingiva | From the implant loading to 36-months of follow-up
  Calibrated probes of 1, 2, 3, 5, 7, and 10 mm will be used to measure the range of keratinized gingiva as the distance from the gingival margin to the mucogingival junction, at the center of the buccal surface. The thickness of the keratinized tissue will be assessed and categorized as thick or thin. This assessment will be based on the transparency of the same periodontal probe through the gingival margin during the probing of the sulcus in the mid-buccal region. If the outline of the underlying periodontal probe could be seen through the gingiva, it was classified as thin (score: 0); otherwise, it was classified as thick (score: 1)